CLINICAL TRIAL: NCT06278233
Title: An Investigation of the Effect of 5 Consecutive Days of Bihemispheric TDCS on Speech Fluency in Individuals With Stuttering
Brief Title: Bihemispheric Transcranial Direct Current Stimulation* on Speech Fluency
Acronym: TDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Feyzanur Ocak, speech therapist, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/85-70
Record Dates: First submitted 2024-02-08; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Stuttering, Adult
Keywords: stuttering; tDCS; non-invasive brain stimulation; speech therapy
MeSH Terms: conditions — Stuttering; Communication Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: In this study, a double-blind, randomized controlled research design from experimental research methods will be applied.
Who Masked: Participant, Outcomes Assessor
Masking Description: One researcher not involved in any aspect of the study will randomize participants to the sham and tDCS study arms using blocked randomization. To ensure blinding, one researcher will record the administration of the tDCS and assessments, while independent speech-language pathologists will monitor the assessment recordings and score the test items.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial direct current stimulation study arm (Experimental): For bi-hemispheric stimulation, the anode will be placed at the intersection of F7 and FC5 and the cathode will be placed at the intersection of F8 and FC6. For all stimulations, the stimulation will be increased for 15 seconds at a dosage of 1 mA (milliampere) for the entire 20 minute session duration and decreased for 15 seconds at the end of the stimulation.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation study arm (No Intervention): In the sham condition, the same electrode placement will be used, during which the current will be increased for 15 seconds, kept at 1 mA for 15 seconds, decreased for 15 seconds and terminated, and the 20 minute session duration will be performed with 45 seconds of real stimulation accompanied by speech with a metronome.

INTERVENTIONS:
Device: Transcranial direct current stimulation — TDCS involves applying a weak electrical current across the head through electrodes placed on the scalp and modulating the resting membrane potential of neurons in the underlying cortex.
  Arms: Transcranial direct current stimulation study arm

SUMMARY:
It will be determined whether bihemispheric stimulation (anodal to the left IFG and cathodal to the right IFG) is used with fluency-facilitating conditions for 5 consecutive days in individuals with stuttering and whether there is a difference in terms of the effects seen in speech fluency compared to the sham condition.

DETAILED DESCRIPTION:
Developmental stuttering is a fluency disorder that can negatively affect many aspects of an individual's life. Recent transcranial direct current stimulation (tDCS) studies with individuals with stuttering show that tDCS shows promise in increasing fluency when used in combination with situations that temporarily increase fluency. In this study, it was aimed to investigate the effect of bi-hemispheric tDCS on fluency in individuals with stuttering for 5 consecutive days. The hypothesis of the study is that bi-hemispheric stimulation, which includes anodal stimulation to the left hemisphere and cathodal stimulation to the right hemisphere, will be effective on reading and speech fluency when performed for 5 consecutive days. Thirty-six adults with developmental stuttering are expected to complete this double-blind, sham-controlled study. Participants will be divided into two groups by blocked randomization and one group will receive sham stimulation for 5 consecutive days and the other group will receive bihemispheric stimulation. Participants in the tDCS group will receive 20 minutes of tDCS stimulation accompanied by metronome-timed speech during the practice sessions. Reading and speaking fluency will be assessed immediately before, immediately after, and one week after the stimulation sessions. Data will be collected using the stuttering severity assessment instrument (SSI-4) Results will be compared both within and between groups in terms of percentage of stuttered syllables, stuttering severity, and evaluation of the speaker's experience of stuttering.

ELIGIBILITY:
Inclusion Criteria:

* developmental stuttering
* age between 18 and 60 years
* right hand dominant

Exclusion Criteria:

* history of seizures, head trauma, hearing problems, cochlear implant, intracranial metal implantation, medications that affects the central nervous system, implanted neurostimulators, cardiac pacemakers, or medication infusion devices
* any speech and language disorder other than developmental stuttering
* neurological or psychiatric disorders, brain surgery, tumours, neurodevelopmental disorders, or attention deficit hyperactivity disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Disfluent syllables | immediately before and immediately after the stimulation on each day of the 5-day intervention, and at 1 week after the end of the intervention.
  change in % disfluent syllables from baseline

SECONDARY OUTCOMES:
Stuttering Severity Instrument- Fourth Edition (SSI-IV) score | immediately before and immediately after the stimulation on each day of the 5-day intervention, and at 1 week after the end of the intervention.
  It measures stuttering severity in the following four areas of speech behavior: (1) frequency, (2) duration, (3) physical concomitants, and (4) naturalness of the individual's speech. Frequency is expressed in percent syllables stuttered and converted to scale scores of 2-18. Duration is timed to the nearest one tenth of a second and converted to scale scores of 2-18. The four types of Physical Concomitants (Distracting Sounds, Facial Grimaces, Head Movements, and Movements of the Extremities) are converted to scale scores of 0-20. Naturalness is ranked on a scale from 1 (Highly Natural Sound Speech) to 9 (Highly Unnatural Sound Speech). Overall naturalness is ranked at the discretion of the clinician. Scaled scores of Frequency, Duration, and Physical Concomitants are added together to derive a Total Score, Percentile Rank, and Severity Equivalent.
The Overall Assessment of the Speaker's Experience of Stuttering (OASES) score | baseline, after the 5-day stimulation and at the 1-week post-intervention time point
  The instrument, which requires approximately 20 min to complete, is organized into four sections: (a) General Information, (b) Reactions to Stuttering, (c) Communication in Daily Situations, and (d) Quality of Life. OASES consists of 100 items, each scored on a Likert scale ranging from 1 to 5. For each item on the OASES, response scales are that higher scores indicate a greater degree of negative impact associated with stuttering and lower scores indicate less negative impact. All impact scores range from a minimum score of 20 (if the speaker answers 1 for every item within a section) up to a maximum of 100 (if the speaker answers 5 for every item within the section).

CONTACTS AND LOCATIONS:
Overall Officials: Feyzanur Ocak, Slp, Principal Investigator — Atlas University; Talat Bulut, Asst. prof., Study Chair — Medipol University; Çağdaş Karsan, Asst. prof., Study Director — Biruni University
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made publicly available with a DOI (digital object identifier) number.
Time Frame: during submission of article
Access Criteria: public and no criteria
URL: http://osf.io

REFERENCES:
- [Background] Yada Y, Tomisato S, Hashimoto RI. Online cathodal transcranial direct current stimulation to the right homologue of Broca's area improves speech fluency in people who stutter. Psychiatry Clin Neurosci. 2019 Feb;73(2):63-69. doi: 10.1111/pcn.12796. Epub 2018 Dec 11. PMID 30379387
- [Background] Garnett EO, Chow HM, Choo AL, Chang SE. Stuttering Severity Modulates Effects of Non-invasive Brain Stimulation in Adults Who Stutter. Front Hum Neurosci. 2019 Nov 21;13:411. doi: 10.3389/fnhum.2019.00411. eCollection 2019. PMID 31824276
- [Result] Chesters J, Mottonen R, Watkins KE. Transcranial direct current stimulation over left inferior frontal cortex improves speech fluency in adults who stutter. Brain. 2018 Apr 1;141(4):1161-1171. doi: 10.1093/brain/awy011. PMID 29394325